CLINICAL TRIAL: NCT03879954
Title: Comparison Between Ultrasound-guided Out-of-plane Internal Jugular Vein and In-plane Supraclavicular Subclavian Vein Catheterization in Intensive Care Unit Patients-a Randomized Trial
Brief Title: US-guided OOP Internal Jugular Vein Vs IP Supraclavicular Subclavian Vein Catheterization in ICU
Acronym: IPSSCVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Trabelsi Becem, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTEM SSCV
Record Dates: First submitted 2019-03-02; First posted 2019-03-19 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Central Venous Catheter

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OOP-IJV (Other): Out of plane inetrnal jugular vein catetherization
  Interventions: Device: Catetherization approach
- IP-SSV (Other): in plane supraclavicular subclavian vein catetherization
  Interventions: Device: Catetherization approach

INTERVENTIONS:
Device: Catetherization approach — Out of plane inetrnal jugular vein Vs in plane supraclavicular subclavian vein catetherization

SUMMARY:
Patients were randomly divided into two groups: ultrasound-guided (US-guided) out-of-plane internal jugular vein (OOP-IJV) and in-plane supraclavicular subclavian vein (IP-SSV) catheterization.

For OOP-IJV cannulation, the transducer was placed to identify IJV in short-axis view. The needle was introduced at an angle of 60° to the skin surface, and advanced under real-time US guidance until visualizing the tip of the needle inside the vein.

For IP-SSV cannulation, a short-axis view of the IJV was obtained first. The probe was slid caudally following the IJV until getting the best long-axis view of the SCV. Using an in-plane approach, the needle was inserted at the base of the transducer at a 30° angle and advanced under the long axis under real-time US guidance targeting the SCV.

DETAILED DESCRIPTION:
Patients were randomly divided into two groups: ultrasound-guided (US-guided) out-of-plane internal jugular vein (OOP-IJV) and in-plane supraclavicular subclavian vein (IP-SSV) catheterization.

For OOP-IJV cannulation, the transducer was placed on transverse position over the patient's neck at the level of the cricoid cartilage to identify IJV and carotid artery (CA) in short-axis view. The vein was then centered on the screen. The skin puncture was made in the center of the US image using a needle attached to a syringe. The needle was introduced at an angle of 60° to the skin surface, perpendicular to the transducer, and advanced under real-time US guidance toward the IJV until visualizing the tip of the needle inside the vein.

For IP-SSV cannulation, a short-axis view of the IJV was obtained first. The probe was slid caudally following the IJV until the junction of the subclavian vein (SCV) and IJV was reached in the supraclavicular fossa. The probe was then turned slightly and tilted anteriorly to get the best long-axis view of the SCV and the brachiocephalic vein (BCV).

Using an in-plane approach, the needle attached to a syringe was inserted at the base of the transducer at a 30° angle and advanced strictly under the long axis of the US probe from lateral to medial. The needle point was then guided under real-time US guidance targeting the SCV.

In both groups, catheterization was done through Seldinger technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit requiring a central venous catheter (CVC)

Exclusion Criteria:

* Major blood coagulation disorders,
* Any thrombotic formations within the vein,
* Congenital or acquired deformity of neck or clavicle
* Cannulation site infection, hematoma and surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
The overall access time | During the venous cannulation procedure
  Time from the ultrasound scanning to the ultrasound confirmation of the correct position of the guidewire into vein.

SECONDARY OUTCOMES:
The guidewire time | During the venous cannulation procedure
  Time from the first skin puncture to the ultrasound confirmation of the correct placement of the guidewire into the vein.
The venous access time | During the venous cannulation procedure
  The time between the first skin puncture and free aspiration of venous blood in the syringe

CONTACTS AND LOCATIONS:
Overall Officials: BEN ALI MECHAAL, PROFESSOR, Study Chair — University Tunis El Manar
Locations (1):
- Mrezga Nabeul Tunisie, Nabeul, Tunisia

REFERENCES:
- [Derived] Trabelsi B, Hajjej Z, Drira D, Yedes A, Labbene I, Ferjani M, Ben Ali M. Comparison of ultrasound-guided internal jugular vein and supraclavicular subclavian vein catheterization in critically ill patients: a prospective, randomized clinical trial. Ann Intensive Care. 2022 Oct 1;12(1):91. doi: 10.1186/s13613-022-01065-x. PMID 36183049